CLINICAL TRIAL: NCT04051034
Title: Heat Therapy and Omega 3 on Metabolic and Cardiovascular Health
Brief Title: Heat Therapy and Omega 3 on Cardio-Metabolic Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Eric Rivas, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2018-1199
Record Dates: First submitted 2019-07-24; First posted 2019-08-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo or Omega 3 supplementation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 supplementation (Experimental): 12 weeks: Active: 1.25 g capsules/ [1.25 g capsule contains min. 750 mg EPA + 250 mg DHA] with heat therapy increasing internal body temperature 1.2C above baseline for 90 min each bout..
  Interventions: Dietary Supplement: Omega 3
- Placebo (Experimental): 12 weeks: Placebo: 1.25 g capsules/ [1.25-gram high oleic safflower oil capsule]with heat therapy increasing internal body temperature 1.2C above baseline for 90 min each bout..
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3 — Active: 1.25 g capsules/420 35-count bottles [1.25 g capsule contains min. 750 mg EPA + 250 mg DHA] and heat therapy, increase internal body temperature 1.2 C above baseline.
  Placebo: 14,700 1.25 g capsules/420 35-count bottles [1.25-gram high oleic safflower oil capsule]
  Other Names: Organic Technologies
  Arms: Omega 3 supplementation
Other: Placebo — Active: 1.25 g capsules [1.25-gram high oleic safflower oil capsule] and heat therapy, increase internal body temperature 1.2 C above baseline.
  Arms: Placebo

SUMMARY:
Currently, controlled studies are lacking which test the benefits of: 1) ω3 PUFA; and 2) heat therapy on improving vascular-metabolic-microbiota health in Hispanic American populations. The investigator's objective is to determine if this modality (heat therapy i.e., warm water immersion, hot tubs) combined with dietary interventions (increased fish and/or fish oil intake) may be feasible treatments to improve cardiovascular risk factors and reduced comorbidities in Hispanic populations.

DETAILED DESCRIPTION:
In a double-blind, placebo-controlled design, participants will be randomized to the following experimental treatments:

1. 4 g omega 3 daily for 12 weeks combined with 6 weeks of heat therapy
2. Placebo pill daily for 12 weeks with 6 weeks of heat therapy (HT)

non-obese healthy will only serve as controls and enroll in placebo and neutral control therapy conditions.

HT will entail 14 consecutive days of 1.5 hours passive heating (increase internal temperature 1.2°C above baseline), followed by 4 weeks of HT, 3 days per week.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30-40,
* fasting glucose 100-125,
* blood pressure 130-139/80-89,
* Hispanic American,
* age 18-65 years

Exclusion Criteria:

* non-Hispanic,
* BMI<30, >40,
* fasting glucose <100, >125,
* blood pressure <130,>139 systolic, >90 diastolic,
* age <18, >65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-20 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic flexibility | Change from baseline to 12 week metabolic flexibility
  Mixed meal tolerance test
Microbiome | Change from baseline to 12 week in the phyla, genus and species of gut bacteria
  Stool microbiome diversity
Short chain fatty acids | Change from baseline to 12 week short chain fatty acids, acetate, propionate, and butyrate (C4).
  Stool Short chain fatty acids
Vascular Health | Change from baseline to 12 week vessel function
  Brachial and skin flow mediated dilation

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Rivas, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF